CLINICAL TRIAL: NCT05880654
Title: IL-39 & IL-35 Gingival Crevicular Fluid Levels in Diabetic Patients With Generalized Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Sandy Hassan, Associate professor oral medicine & periodontology departement, Fayoum University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #REC-FDBSU/06102022-02/HS
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Generalized Periodontal Disease, AVDC Stage 3
Keywords: Periodontitis & Diabetes mellitus
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus | interventions — Tooth Exfoliation

STUDY DESIGN:
Intervention Model Description: Chronic periodontitis group chronic periodontitis with diabetes control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Systemically healthy periodontitis (Active Comparator): Non Surgical Periodontal therapy ( Scaling & Root planning)
  Interventions: Procedure: Scaling & root planning
- Diabetic & Periodontitis (Active Comparator): Non surgical periodontal therapy ( scaling & root planning)
  Interventions: Procedure: Scaling & root planning
- Control (No Intervention): Healthy group with neither Diabetes nor Periodontitis

INTERVENTIONS:
Procedure: Scaling & root planning — Non Surgical periodontal therapy
  Arms: Diabetic & Periodontitis; Systemically healthy periodontitis

SUMMARY:
The sudy was aiming to assess and compare GCF levels of IL-39 & IL-35 in gingival crevicular fluid and to correlate the relationship between different patient groups before and after non-surgical therapy.

DETAILED DESCRIPTION:
Methodology:

Group I (Periodontitis Group): 19 patients suffering from generalized periodontitis with T2DM age range, 35-50 years.

Group II (Periodontitis Group): 19 patients suffering from generalized periodontitis & systemically healthy, age range: 35-50 years.

Group III (Control group): 19 Periodontally and systemically healthy volunteers who served as control subjects age range: 30-45 years.

Periodontitis participants will be collected from the outpatient clinic of oral medicine and periodontology departments in Fayoum, Beni-Swief and Ahram-Candian universities. The periodontitis included subjects will be diagnosed according to the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions (Tonetti, MS, Greenwell, H, Kornman, KS. Staging and grading of periodontitis: framework and proposal of a new classification and case definition. J Periodontol.; 89( Suppl 1): S159- S172, 2018.)

Diabetic patients will be enrolled in this study according to the criteria of American Diabetes Association. (American Diabetes Association. (2) Classification and diagnosis of diabetes. Diabetes Care 38: S8-S16, 2015.)

The control group will be selected from healthy subjects who attended the restorative dental clinic and has apparently clinically healthy gingiva.

Micropipettes will be used for collection of GCF samples for control group and periodontitis patients before & after periodontal treatment.

A complete mouth non-surgical periodontal therapy will be carried out for both periodontitis groups

The levels of IL-35 in the GCF samples were assessed using an ELISA kit following the guidelines by the manufacturer.

ELIGIBILITY:
Inclusion Criteria Stage III Grade C Generalized periodontitis with diabetes Stage III grade B Generalized periodontitis in systemic healthy subjects

Exclusion Criteria:

1. Patients treated with any type of medications and/ or antibiotics during the past 3 months,
2. Pregnancy
3. Lactation
4. Receiving professional periodontal treatment during the past 6 months
5. Current or former smokers

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
GCF levels of IL-39 & IL35 | 3 months
  Gingival crevicular fluid levels of IL-39 & IL-35 in healthy & diabetic patients with periodontitis
Effect of SRP on GCF levels of IL-39 & IL35 | 3 MONTHS
  Gingival crevicular fluid levels of IL-39 & IL-35 in healthy & diabetic patients with periodontitis after Scaling & root planning

CONTACTS AND LOCATIONS:
Overall Officials: sandy Hassan, ass.prof, Principal Investigator — associate professor
Locations (2):
- Egypt (2):
  - Sandy hassan, Cairo, Virginia
  - Sandy hassan shaaban, Cairo